CLINICAL TRIAL: NCT00062517
Title: Generalized Anxiety Disorder and Social Anxiety Disorder: Their Impact on the Processing of Social Emotional Information and Instrumental Learning
Brief Title: Generalized Anxiety Disorder and Social Anxiety Disorder: Their Impact on the Processing of Information and Learning
Status: Completed | Type: Observational
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 030185; 03-M-0185
Record Dates: First submitted 2003-06-06; First posted 2003-06-09 (Estimated); Last update posted 2017-10-06 (Actual); Status verified 2016-09-21

CONDITIONS: Anxiety Disorders
Keywords: Amygdala; Generalized Anxiety Disorder; Anxiety Disorder; GAD; Social Anxiety Disorder; SAD
MeSH Terms: conditions — Anxiety Disorders; Generalized Anxiety Disorder; Phobia, Social

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
The purpose of this study is to increase researchers understanding of the biological basis of generalized anxiety disorder and social anxiety disorder. They will investigate how the brain activity associated with specific thoughts and feelings may play a role in these anxiety disorders. This knowledge will be used to design interventions to help those with these illnesses.

To qualify for this study, participants must be evaluated via an initial telephone screening interview and material sent through the mail.

Participants will then be required to make three visits to NIH. During the first visit, they will be asked questions about their general mood, degree of nervousness, thinking skills, and behavior. They will undergo a thorough physical exam, including an EKG, blood work, urinalysis, and a pregnancy test for women of childbearing potential. During the second visit, participants will spend about 2.5 hours doing various tasks while sitting and looking at a computer screen. These tasks will guide them to experience specific kinds of thoughts and emotions. Researchers will attach electrodes to the participants hands to monitor the amount of electricity conducted by the skin. The third visit will be similar to the second visit, but participants will perform the tasks while lying in a MRI scanner.

Participants will be compensated up to $400 for their involvement in this study.

DETAILED DESCRIPTION:
There have been suggestions that the threshold for amygdala activity is lower in individuals with anxiety disorders than in healthy individuals. However, despite it's immediate plausibility, there have been relatively few tests of this hypothesis. Specifically, there have been very few explorations of the performance of patients with anxiety disorders on measures known to implicate the amygdala.

Although the high co-morbidity of Generalized Anxiety Disorder (GAD) and Social Anxiety Disorder (SAD) complicates the issue, the fact that the disorders doubly dissociate suggests that they are due to dysfunctional activity in separable neurocognitive systems. We would suggest that the hyper-responsive amygdala hypothesis is more likely to be linked to the explanation of GAD. In contrast, SAD may be due to reduced activation thresholds for units in a system that responds to social threat and which recruits lateral orbital frontal cortex. Thus, the current project will determine the performance of patients with GAD and SAD on measures in which the amygdala is known to play a role and also measures that recruit lateral orbital frontal cortex and the system for social response reversal. In addition, two proposed neuro-imaging studies will directly assess neural responses in these two systems in both patient populations. The project should provide clear data that will constrain future theorizing on the pathology implicated in these two disorders.

ELIGIBILITY:
* INCLUSION CRITERIA:

Age: Participants will be males and females, 18-50 years of age.

IQ: IQ, as measured by 4 subscales from the Wechsler Adult Intelligence Scale-Revised (WAIS-R), must be > 80.

Medication status: No regular use of psychotropic medication within 2 weeks of the study (or fluoxetine within 8 weeks of the study). No regular use of any benzodiazepine. We intend to identify patients whose GAD/SAD is currently untreated.

EXCLUSION CRITERIA:

Because factors such as psychiatric disease, or CNS disease, can influence functional brain activity, and pregnancy precludes participation in fMRI studies, these factors are exclusionary.

1. Psychiatric history: Participants will be assessed using DSM-IV criteria via standardized psychiatric interviews conducted by trained examiners (i.e., SCID). Any current suicidal ideation will be exclusionary.

   1. Healthy comparison individuals (Group 1): All participants will be free of any current psychiatric disorder as well as lifetime history of psychosis, pervasive developmental disorder, major affective disorder, panic disorder, obsessive compulsive disorder, conduct disorder, ADHD, anorexia.
   2. Patients with GAD (Group 2): Any history of an axis I diagnosis excluding SAD but not including adjustment disorder, simple phobia or dysthymia is exclusionary. There must be no current mood disoder (MD) though patients with past MD, which occurred after the onset of GAD, will be admitted to the study. We recognize the difficulty of recruiting patients with GAD without co-morbid SAD and will therefore allow patients who are comorbid into the study in this group. We have faced difficulties with our studies of children with psychopathic tendencies where, although it is possible to identify populations who only meet criteria for ADHD most children who meet criteria for psychopathic tendencies are co-morbid for ADHD. We will adopt a similar strategy to our work with children; i.e., in contrasts of patients with GAD with comparison individuals, we will use SAD symptomatology as a covariate to reduce, and evaluate, the impact of pathology associated with SAD on the data.
   3. Patients with SAD (Group 3): Any current history of an axis I diagnosis including GAD, but excluding adjustment disorder, simple phobia or dysthymia is exclusionary. There must be no current mood disorder (MD) though patients with past MD, which occurred after the onset of SAD, will be admitted to the study.
2. History of Drug Abuse: Axis I diagnoses of substance use disorders will be exclusionary.
3. Severe acute and chronic medical illnesses.
4. CNS disease: History of brain abnormalities (e.g., neoplasms, subarachnoid cysts), cerebrovascular disease, infectious disease (e.g., abscess), or other neurological disease, or history of head trauma (defined as loss of consciousness > 3 min).
5. Metal or electronic objects: Metal plates, certain types of dental braces, cardiac pacemakers, etc., that are sensitive to electromagnetic fields contraindicate MRI scans.
6. Claustrophobia: Participants will be questioned about potential discomfort in being in an enclosed space, such as an MRI scanner.
7. Pregnancy status: Because of the potential effects of hormonal changes on brain function as well as the unknown effects of electromagnetic field on the fetus, known pregnancy is an exclusion criterion.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 497 (Actual)
Dates: Start 2003-06-05; Study Completion 2016-09-21

PRIMARY OUTCOMES:
Association of GAD/SAD with amygdala act | Ongoing

CONTACTS AND LOCATIONS:
Overall Officials: Karina S Peschardt, Ph.D., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Adolphs R, Tranel D, Hamann S, Young AW, Calder AJ, Phelps EA, Anderson A, Lee GP, Damasio AR. Recognition of facial emotion in nine individuals with bilateral amygdala damage. Neuropsychologia. 1999 Sep;37(10):1111-7. doi: 10.1016/s0028-3932(99)00039-1. PMID 10509833
- [Background] Ambrogi Lorenzini CG, Baldi E, Bucherelli C, Sacchetti B, Tassoni G. Neural topography and chronology of memory consolidation: a review of functional inactivation findings. Neurobiol Learn Mem. 1999 Jan;71(1):1-18. doi: 10.1006/nlme.1998.3865. PMID 9889069
- [Background] Bechara A, Damasio H, Damasio AR, Lee GP. Different contributions of the human amygdala and ventromedial prefrontal cortex to decision-making. J Neurosci. 1999 Jul 1;19(13):5473-81. doi: 10.1523/JNEUROSCI.19-13-05473.1999. PMID 10377356